CLINICAL TRIAL: NCT04329845
Title: Myth and Facts About the Evolving Role of Laparoscopic Splenectomy in Isolated High Grades Splenic Injuries in Hemodynamically Stable Patients With Blunt Abdominal Trauma .Randomized Controlled Trials
Brief Title: Laparoscopic Splenectomy in Isolated High Grades Splenic Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, assistant professour, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: zagazig 6
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Laparoscopic Surgery
Keywords: laparoscopy; laparotomy; non-penetrating; splenectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open splenectomy for splenic injury in trauma (Active Comparator): open splenectomy as a technique for removal of the spleen in case of injury to spleen
  Interventions: Procedure: open splenectomy
- laparoscopic splenectomy for splenic injury in trauma (Active Comparator): laparoscopic splenectomy as a technique for removal of the spleen in case of injury to spleen
  Interventions: Procedure: laparoscopic splenectomy for splenic injury in trauma

INTERVENTIONS:
Procedure: open splenectomy — open splenectomy for treatment of splenic injury
  Arms: open splenectomy for splenic injury in trauma
Procedure: laparoscopic splenectomy for splenic injury in trauma — laparoscopy as a technique for removal of the spleen in injury
  Arms: laparoscopic splenectomy for splenic injury in trauma

SUMMARY:
Background: Trauma laparoscopic splenectomy has no defined reasons. Compared trauma patient characteristics and results with laparoscopic and open splenectomies.

Methods: Patients aged 15 or older with blunt splenic injuries from January 2012 to July 2017 needed splenectomy. Demographics, splenic damage grade, approach (open or laparoscopic), surgery duration, intra-operative blood loss, transfusions, hospital stay, complications, and death were variables.

DETAILED DESCRIPTION:
The spleen might be injured in left lower chest or upper abdomen trauma. Rib cage, diaphragm, pancreas, and bowel injuries may occur with splenic injuries. Hemodynamic instability, a rising heart rate, and low blood pressure are symptoms of damage, however the mechanism of injury requires a high index of suspicion.

ELIGIBILITY:
Inclusion Criteria:

* • At least 15 years old.

  * Male and female (not pregnant) patients; • Sonar and CT scans before surgery showed single splenic damage;

Exclusion Criteria:

* • Other damage to the abdomen, thorax, or nerves were found before surgery.

  * good use of non-surgical treatment or embolization
  * Woman who is pregnant.
  * Splenic cuts that go deep.
  * Previous surgery in the upper abdomen using a laparoscopic method. • Other injuries to the abdomen found during surgery, such as liver, intestine, or bladder injuries.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
mortality | 1.5 years
  during operation or immediate postoperative

SECONDARY OUTCOMES:
intraoperative complications | 5 years
  intraoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: tamer A. alnaimy, MD, Principal Investigator — Zagazig University

IPD SHARING:
Plan to Share IPD: No